CLINICAL TRIAL: NCT02559102
Title: Dexmedetomidine Sedation Versus General Anaesthesia for Inguinal Hernia Surgery on Peri-operative Outcomes and Neurocognitive Development in Infants: A Randomized Controlled Trial
Brief Title: Dexmedetomidine Sedation Versus General Anaesthesia for Inguinal Hernia Surgery in Infants
Acronym: DEGA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Singhealth Foundation (Other Government); Institute for Human Development and Potential (IHDP), Singapore (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHF/CTG055/2014
Record Dates: First submitted 2015-08-04; First posted 2015-09-24 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2017-03

CONDITIONS: Neurodevelopmental Disorder; Bilateral Inguinal Hernia
Keywords: Dexmedetomidine sedation; General anaesthesia; Neurodevelopment; Infants; Neonates
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Gases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dex Group (Experimental): Intravenous dexmedetomidine sedation prior to single shot caudal anaesthesia and maintenance infusion of dexmedetomidine during bilateral inguinal hernia surgery.
  Interventions: Drug: Dexmedetomidine sedation; Procedure: Caudal anaesthesia; Procedure: Inguinal hernia surgery
- GA Group (Active Comparator): General sevoflurane anaesthesia with endotracheal intubation and single shot caudal anaesthesia for inguinal hernia surgery. This is currently the standard anaesthetic technique for bilateral inguinal hernia surgery in neonates and infants in KKH.
  Interventions: Drug: General sevoflurane anaesthesia; Procedure: Caudal anaesthesia; Procedure: Inguinal hernia surgery

INTERVENTIONS:
Drug: Dexmedetomidine sedation — Patients receive dexmedetomidine sedation
  Other Names: Dex
  Arms: Dex Group
Drug: General sevoflurane anaesthesia — Patients receive general sevoflurane anaesthesia with endotracheal intubation
  Other Names: Gas
  Arms: GA Group
Procedure: Caudal anaesthesia — single shot caudal anaesthesia
  Other Names: Caudal
Procedure: Inguinal hernia surgery — Infant inguinal hernia repair.
  Other Names: Inguinal herniotomy

SUMMARY:
This is a prospective randomized controlled trial comparing dexmedetomidine sedation with caudal anaesthesia, and general sevoflurane anaesthesia with caudal anaesthesia for inguinal herniotomies in neonates and infants below 3 months of age.

The investigators will compare the efficacy and adverse events associated with each of these techniques and neurodevelopmental outcomes of the infants in each group at 6 months and 2 years of age.

DETAILED DESCRIPTION:
Several epidemiologic studies have suggested that children exposed to general anaesthesia (GA) in early childhood may be at increased risk of subsequent learning disabilities and behavioural problems. Animal studies have shown that exposure to GA agents during critical neuro-developmental windows induces neuronal apoptosis. All commonly used anaesthetic agents induce neurotoxicity with the exception of dexmedetomidine, a highly specific alpha-2 agonist which has been shown to be neuroprotective.

GA is the current standard of care for inguinal hernia repair in infants at KKH. The investigators recently demonstrated that dexmedetomidine sedation with caudal block is a feasible alternative for inguinal hernia repair in infants below 3 months of age. This prospective randomized controlled trial will compare the early and long-term outcomes of infants following inguinal hernia surgery using dexmedetomidine sedation with caudal block versus GA with caudal block.

This study aims:

1. To compare the neurodevelopment at 6 months and 2years, of infants randomized to dexmedetomidine sedation with caudal block with those randomized to GA with caudal block for inguinal hernia surgery before 3 months of age.
2. To compare the efficacy of dexmedetomidine sedation with caudal block versus GA with caudal block for inguinal hernia surgery, in terms of duration of anaesthesia, duration of surgery and surgeon's satisfaction with intraoperative conditions.

ELIGIBILITY:
Inclusion Criteria:

* Infants below 3 months of age ( corrected age 54 weeks) presenting for elective inguinal hernia repair in KKH.

Exclusion Criteria:

* History of prematurity younger than 28 weeks gestation,
* Requirement for CPAP greater than 6 cmH20 at time of surgery
* Significant cardiac pathology or cardiac conduction defects
* Unusually large hernia sacs
* Any contraindication for caudal anesthesia
* Surgeon refusal on account of anticipated prolonged or difficult surgery.

Ages: 34 Weeks to 54 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2015-07; Primary Completion 2020-07-20 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Deferred Imitation scores at 6 months | 6 months
  Deferred imitation, test of declarative memory. Infants are assessed when first shown the "target" actions (DF1) and again on how well they reproduce the actions (DF2).

SECONDARY OUTCOMES:
Bayley scores at 2 years | 2 years
  Bayleys scales of Infant Development version III

OTHER OUTCOMES:
Surgical success rate | 4 hours
  Success rate of surgery with assigned technique, without requiring further adjuvants.
Peri-operative apnea episodes | 24 hours
  Number of episodes of apnea intra-operatively, in PACU, and in ward.
Peri-operative bradycardic episodes | 24 hours
  Number of episodes of bradycardia intra-operatively, in PACU, and in ward.

CONTACTS AND LOCATIONS:
Overall Officials: Choon L Bong, MBChB FRCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

REFERENCES:
- [Background] Jevtovic-Todorovic V, Hartman RE, Izumi Y, Benshoff ND, Dikranian K, Zorumski CF, Olney JW, Wozniak DF. Early exposure to common anesthetic agents causes widespread neurodegeneration in the developing rat brain and persistent learning deficits. J Neurosci. 2003 Feb 1;23(3):876-82. doi: 10.1523/JNEUROSCI.23-03-00876.2003. PMID 12574416
- [Background] Sanders RD, Sun P, Patel S, Li M, Maze M, Ma D. Dexmedetomidine provides cortical neuroprotection: impact on anaesthetic-induced neuroapoptosis in the rat developing brain. Acta Anaesthesiol Scand. 2010 Jul;54(6):710-6. doi: 10.1111/j.1399-6576.2009.02177.x. Epub 2009 Dec 9. PMID 20003127
- [Background] Mahmoud M, Mason KP. Dexmedetomidine: review, update, and future considerations of paediatric perioperative and periprocedural applications and limitations. Br J Anaesth. 2015 Aug;115(2):171-82. doi: 10.1093/bja/aev226. PMID 26170346
- [Derived] Bong CL, Tan J, Lim S, Low Y, Sim SW, Rajadurai VS, Khoo PC, Allen J, Meaney M, Koh WP. Randomised controlled trial of dexmedetomidine sedation vs general anaesthesia for inguinal hernia surgery on perioperative outcomes in infants. Br J Anaesth. 2019 May;122(5):662-670. doi: 10.1016/j.bja.2018.12.027. Epub 2019 Mar 7. PMID 30916007